CLINICAL TRIAL: NCT05494281
Title: Serratus Anterior Plane Block to Prevent Chronic Pain in Breast Cancer Surgery: A Randomized Controlled Trial
Brief Title: Serratus Anterior Plane Block to Prevent Chronic Postoperative Pain in Breast Cancer
Acronym: USB22
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Moroccan Society of Surgery (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: USB_22 Trial
Record Dates: First submitted 2022-08-06; First posted 2022-08-09 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Breast Neoplasms; Pain, Postoperative; Pain, Chronic; Post-Mastectomy Chronic Pain Syndrome
MeSH Terms: conditions — Breast Neoplasms; Pain, Postoperative; Chronic Pain | interventions — Anesthetics, Local; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Experimental)
  Interventions: Procedure: Serratus Anterior Plane Block with saline solution
- Serratus anterior plane block (Experimental)
  Interventions: Procedure: Serratus Anterior Plane Block with local anesthetic

INTERVENTIONS:
Procedure: Serratus Anterior Plane Block with local anesthetic — A deep analgesic block of the Serratus anterior plane block (SAPB) type by echo-guided lateral approach will be performed by An 8-13 Mhz high frequency linear ultrasound probe witch will be located cranio-caudally, transversely to the 3rd and 4th intercostal space on the mid-axillary line while patients are supine with the ipsilateral upper limb raised to 90°.
  Once the landmark anatomical structures have been identified (upper rib, lower rib, pleural line, Serratus muscle, superficial structures), the puncture will begin Under aseptic conditions, an 80 mm 22 gauge needle will be inserted into the "in-plane" view of the ultrasound probe. When the needle has reached the plane under Serratus between the Serratus muscle and the intercostal muscle opposite the lower edge of the upper rib, 30 ml of 1% Lidocaine will be administered.
  Arms: Serratus anterior plane block
Procedure: Serratus Anterior Plane Block with saline solution — A deep analgesic block of the Serratus anterior plane block (SAPB) type by echo-guided lateral approach will be performed by An 8-13 Mhz high frequency linear ultrasound probe witch will be located cranio-caudally, transversely to the 3rd and 4th intercostal space on the mid-axillary line while patients are supine with the ipsilateral upper limb raised to 90°.
  Once the landmark anatomical structures have been identified (upper rib, lower rib, pleural line, Serratus muscle, superficial structures), the puncture will begin Under aseptic conditions, an 80 mm 22 gauge needle will be inserted into the "in-plane" view of the ultrasound probe. When the needle has reached the plane under Serratus between the Serratus muscle and the intercostal muscle opposite the lower edge of the upper rib, 30 ml of saline solution
  Arms: Placebo

SUMMARY:
Chronic postoperative pain (CPP) remains a disturbing and obscure clinical problem.

The hypothesis of this trial is that a peripheral block of the serratus anterior plane block type preoperatively after a modified radical mastectomy makes it possible to reduce the intensity and incidence of chronic post-surgical pain in breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Having an age greater than or equal to 18 years and less than 70 years
* Having given written consent for participation in the study and the use of personal and medical data
* Having a physical status of class I, II or III of the American Society of Anesthesiologists

Exclusion Criteria:

* Patients who expressed their refusal to participate in the study
* Patients unable to express their non-objection to participation in the study
* American Society of Anesthesiologists class > III patients
* Known allergy to local anesthetics
* A contraindication to performing a peripheral nerve block (such as an acquired, constitutional or drug clotting disorder or infection at the nerve block injection site)
* Morbid obesity (body mass index greater than 40 kg/m²)
* Chronic use of opioids
* Inability to use the patient controlled analgesia device
* The existence of preoperative pain
* History of neuropathy or neurological pathology
* The existence of catastrophism or anxiety diagnosed preoperatively

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women Having to undergo an elective unilateral modified total mastectomy with dissection of the axillary lymph nodes (modified Patey procedure) for curative purposes for oncological pathology of the breast, performed in the operating room of the Gyneco-mammary center of INO, without breast reconstruction
Enrollment: 94 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Chronic postoperative pain at 3 months | 3 months after surgery
  A question will be asked to patients : "Throughout our lives, most have had pain (like headaches, sprains and toothaches). Have you had pain other than these types of pain on a daily basis since your surgery? " The answer "yes" or "no" will determine the outcome
chronic postoperative pain intensity | 3 months after surgery
  Pain intensity of patients was evaluated by Numerical Rating Scale, rating from 0 (no pain) to 10 (extreme pain) in order to evaluate the effect of Serratus Anterior Plane Block in preventing chronic pain

SECONDARY OUTCOMES:
Chronic Pain intensity and quality | 3 months after surgery
  Pain intensity of patients was evaluated by Arabic version of Brief pain inventory
Neuropathic pain screening | 3 months after surgery
  Neuropathic pain will be screened by "Douleur Neuropathique 4" score
Morphine consumption | 0-24 hours after operation
  Morphine rescue dose for extra need of analgesic

CONTACTS AND LOCATIONS:
Overall Officials: Abdelilah GHANNAM, MD, Study Director — Mohammed V University in Rabat
Locations (1):
- Anesthesia & Critical care department - National Institut of Oncology in Rabat. Ibn Sina teaching Hospital. Mohammed V university of Rabat, Rabat, Morocco

IPD SHARING:
Plan to Share IPD: No